CLINICAL TRIAL: NCT06880744
Title: Phase 3b, Multicenter, Randomized, Open-Label Study of Risankizumab Compared to Vedolizumab for the Treatment of Adult Subjects With Moderate to Severe Ulcerative Colitis Who Are Naïve to Targeted Therapies
Brief Title: A Study to Assess the Change in Disease Activity in Adult Participants With Moderate to Severe Ulcerative Colitis Treated With Risankizumab Compared to Vedolizumab
Acronym: REVAMP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-540
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — risankizumab; vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab Group (Active Comparator): An induction dose of risankizumab intravenous (IV) will be administered at Baseline and Weeks 4 and 8. Starting at Week 12, participants will then receive either a lower or higher subcutaneous (SC) risankizumab maintenance dose, followed by the same dose every 8 weeks with the last dose at Week 44.
  Interventions: Drug: Risankizumab
- Vedolizumab Group (Active Comparator): Vedolizumab IV will be administered at Baseline, Weeks 2 and 6, and every 8 weeks with the last dose of vedolizumab IV at Week 46.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) Infusion
  Arms: Risankizumab Group
Drug: Risankizumab — Subcutaneous (SC) injection
  Arms: Risankizumab Group
Drug: Vedolizumab — Intravenous (IV) infusion
  Arms: Vedolizumab Group

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine).This study will evaluate how safe and effective risankizumab is compared to vedolizumab in treating adult participants with moderate to severe UC who are naive to targeted therapies (TaTs).

Risankizumab and vedolizumab are approved medications for moderate to severe UC in multiple countries. Participants who meet the eligibility criteria will be randomized in a 1:1 ratio to receive open label risankizumab or vedolizumab. Approximately 530 adult participants with moderate to severe UC who are naïve to targeted therapies (TaTs) will be enrolled at 285 sites worldwide.

For participants randomized to risankizumab, drug will be administered intravenous(IV) during the induction period followed by subcutaneous injection during the maintenance period. Participants randomized to vedolizumab will receive drug IV throughout the study.

The duration of the study is approximately 69 weeks for participants randomized to risankizumab and 71 weeks for participants randomized to vedolizumab. This includes up to a 35-day screening period followed by a treatment period of 44 weeks for risankizumab and 46 weeks for vedolizumab.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular outpatient visits during the study. The effect and safety of the treatment will be checked by medical assessments, evaluation of side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant has confirmed diagnosis of Ulcerative Colitis (UC) for at least 3 months prior to Baseline.
* Participant has active UC with an modified Mayo Score (mMS) of 5 to 9 points and endoscopic subscore of 2 to 3 (confirmed by central reader).
* Participant has demonstrated intolerance or inadequate response to one or more of the following categories of drugs: aminosalicylates, oral locally acting steroids, systemic steroids (prednisone or equivalent), and immunomodulators.

Exclusion Criteria:

* Participant has received any targeted therapies (TaTs) for UC, including but not limited to infliximab, etanercept, adalimumab, natalizumab, golimumab, ozanimod, ustekinumab, etrolizumab, vedolizumab, tofacitinib, filgotinib, etrasimod, guselkumab, mirikizumab, upadacitinib, and risankizumab.
* Participant with a current diagnosis of Crohn's disease (CD) or Irritable Bowel Disease (IBD)-unclassified or a history of radiation colitis or ischemic colitis.
* Currently known complications of UC such as: fulminant colitis and/or toxic megacolon, acute severe UC, previous colectomy (total or subtotal), or any other manifestation that might require surgery while in the study
* Active systemic infection/clinically important infection during the last 2 weeks prior to Baseline Visit as assessed by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Risankizumab Group Participants Achieving Endoscopic Improvement As Compared to The Vedolizumab Group | At Week 48
  Endoscopic improvement is defined as endoscopy subscore of 0 or 1. Endoscopies assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).

SECONDARY OUTCOMES:
Percentage of Risankizumab Group Participants who Achieve Clinical Remission As Compared to The Vedolizumab Group Per Modified Mayo Score (mMS) | At Week 48
  Clinical remission on the mMS is defined as Endoscopy subscore = 0 or 1, AND Rectal bleeding subscore = 0, AND Stool frequency subscore <= 1, AND not greater than baseline. The mMS is a composite score of UC disease activity based on the following 3 subscores: SFS, scored from 0 (normal number of stools) to 3 (5 or more stools more than normal); RBS, scored from 0 (no blood seen) to 3 (blood alone passed); ESS, scored from 0 (normal appearance of mucosa) to 3 (severe disease [spontaneous bleeding, ulceration]). The overall mMS ranges from 0 to 9 with higher scores representing more severe disease. The number of responders is calculated based on the total number of participants and estimated response rate, rounding to a nearest whole integer.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (262):
- United States (74):
  - Gastro Health Research - St. Vincent'S East /ID# 275089, Birmingham, Alabama
  - Digestive Health Specialists /ID# 274785, Dothan, Alabama
  - East View Medical Research /ID# 276222, Mobile, Alabama
  - Arizona Health Research /ID# 274366, Chandler, Arizona
  - UC San Diego Health System /ID# 273538, La Jolla, California
  - Gastro Care Institute /ID# 274873, Lancaster, California
  - UCLA Health - Digestive Health & Nutrition Clinic /ID# 274827, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian /ID# 274364, Newport Beach, California
  - California Medical Research Associates /ID# 274787, Northridge, California
  - uc davis medical center - patient support services building /ID# 274251, Sacramento, California
  - Clinical Applications Laboratories - San Diego - 3rd Avenue /ID# 273527, San Diego, California
  - Danbury Hospital, Western Connecticut Health Network /ID# 275277, Danbury, Connecticut
  - Novum Research /ID# 273587, Clermont, Florida
  - Hillcrest Medical Research /ID# 273593, DeLand, Florida
  - Florida Research Institute /ID# 275196, Lakewood Rch, Florida
  - Sanchez Clinical Research /ID# 273727, Miami, Florida
  - Medical Professional Clinical Research /ID# 275208, Miami, Florida
  - Sarkis Clinical Trials - Ocala /ID# 273595, Ocala, Florida
  - Endoscopic Research, Inc. /ID# 273548, Orlando, Florida
  - Digestive And Liver Center Of Florida - Orlando /ID# 276432, Orlando, Florida
  - Emory University School Of Medicine - Atlanta /ID# 273522, Atlanta, Georgia
  - Gi Alliance - Glenview /ID# 274270, Glenview, Illinois
  - Illinois Gastroenterology Group /ID# 274280, Gurnee, Illinois
  - Southwest Gastroenterology - Oak Lawn /ID# 273596, Oak Lawn, Illinois
  - OSF St. Francis Medical Center /ID# 274391, Peoria, Illinois
  - Springfield Clinic Main Campus /ID# 273547, Springfield, Illinois
  - Gastroenterology Health Partners /ID# 276434, New Albany, Indiana
  - Iowa Digestive Disease Center - Clive /ID# 274558, Clive, Iowa
  - Cotton O'Neil Digestive Health Center /ID# 274394, Topeka, Kansas
  - Gastroenterology Health Partners, PLLC /ID# 276441, Louisville, Kentucky
  - Tandem Clinical Research - Houma /ID# 274562, Houma, Louisiana
  - Metropolitan Gastroenterology Associates - Metairie /ID# 274282, Metairie, Louisiana
  - Pinnacle Gastroenterology /ID# 274991, Shreveport, Louisiana
  - Louisiana Research Center, LLC /ID# 276443, Shreveport, Louisiana
  - Velocity Clinical Research, Rockville /ID# 273599, Rockville, Maryland
  - Brigham & Womens Hospital /ID# 275266, Boston, Massachusetts
  - Lucida Clinical Trials /ID# 275235, New Bedford, Massachusetts
  - Huron Gastroenterology /ID# 274998, Ann Arbor, Michigan
  - Mayo Clinic-Rochester /ID# 273606, Rochester, Minnesota
  - Gi Associates - Gia And Endoscopy Center - Flowood /ID# 274285, Flowood, Mississippi
  - Delta Gastroenterology & Endoscopy Center /ID# 275005, Southaven, Mississippi
  - Columbia University Medical Center /ID# 273518, New York, New York
  - New York Gastroenterology Associates - Upper East Side /ID# 273520, New York, New York
  - Gastroenterology Group of Rochester /ID# 274283, Rochester, New York
  - Digestive Health Partners - Biltmore Office /ID# 273594, Asheville, North Carolina
  - Atrium Health - Morehead /ID# 274245, Charlotte, North Carolina
  - Charlotte Gastroenterology And Hepatology - Randolph Road /ID# 274553, Charlotte, North Carolina
  - Carolina Digestive Diseases And Endoscopy Center /ID# 274256, Greenville, North Carolina
  - Digestive Disease Consultants - Brunswick /ID# 276445, Brunswick, Ohio
  - Gastro Health /ID# 275082, Cincinnati, Ohio
  - University Of Cincinnati Medical Center /ID# 273524, Cincinnati, Ohio
  - The Ohio State University - Wexner Medical Center /ID# 274743, Columbus, Ohio
  - Dayton Gastroenterology, Inc /ID# 273528, Dayton, Ohio
  - Digestive Disease Associates, LTD - Wyomissing /ID# 273603, Wyomissing, Pennsylvania
  - Gastroenterology Associates of Orangeburg /ID# 274559, Orangeburg, South Carolina
  - Gastro One - Walnut Run Road /ID# 273551, Cordova, Tennessee
  - Skyline Gastroenterology of West Tennessee /ID# 276461, Jackson, Tennessee
  - GI associates of Northeast Tennessee /ID# 273758, Johnson City, Tennessee
  - Tri-Cities Gastroenterology /ID# 275067, Kingsport, Tennessee
  - Gastrointestinal Associates - Knoxville - Dowell Springs Boulevard /ID# 276447, Knoxville, Tennessee
  - Quality Medical Research /ID# 273733, Nashville, Tennessee
  - Amel Med /ID# 276439, Georgetown, Texas
  - Digestive & Liver Disease Consultants /ID# 276454, Houston, Texas
  - Katy Integrative Gastroenterology /ID# 274645, Katy, Texas
  - Caprock Gastro Research - Lubbock - 80th Street /ID# 273778, Lubbock, Texas
  - GI Alliance: Mansfield /ID# 274272, Mansfield, Texas
  - Linq Research /ID# 274917, Pearland, Texas
  - Tyler Research Institute, LLC /ID# 273585, Tyler, Texas
  - Care Access - Ogden /ID# 274361, Ogden, Utah
  - Gastroenterology Associates Of Tidewater - Chesapeake /ID# 276440, Chesapeake, Virginia
  - Emeritas Research Group /ID# 276457, Lansdowne Town Center, Virginia
  - Gi Alliance - Bellevue /ID# 274264, Bellevue, Washington
  - Virginia Mason Hospital & Medical Center /ID# 274810, Seattle, Washington
  - Washington Gastroenterology - Tacoma /ID# 274551, Tacoma, Washington
- Austria (5):
  - Medizinische Universitaet Graz /ID# 274428, Graz, Styria
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 274318, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 274172, Wels, Upper Austria
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 273611, Salzburg
  - Medizinische Universitaet Wien /ID# 273612, Vienna
- Bulgaria (6):
  - Hospital Tsaritsa Yoanna /ID# 274723, Sofiya, Sofia
  - Umhat Sveti Ivan Rilsky /ID# 274794, Sofiya, Sofia
  - Acibadem City Clinic UMHAT Mladost /ID# 274804, Sofiya, Sofia
  - Umbal Kaspela /ID# 274721, Plovdiv
  - MHAT Knyaginya Klementina /ID# 274722, Sofia
  - Mhat Doverie /ID# 274798, Sofia
- Canada (9):
  - University Of Calgary - Health Sciences Centre /ID# 274237, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institute /ID# 274239, Edmonton, Alberta
  - South Edmonton Gastroenterology /ID# 274184, Edmonton, Alberta
  - Barrie GI Associates /ID# 275211, Barrie, Ontario
  - Brampton Gastroenterology Inc /Id# 276187, Brampton, Ontario
  - GNRR Digestive Clinics and Research Center Inc. /ID# 275820, Brampton, Ontario
  - The Oakville Endoscopy Centre /ID# 275213, Oakville, Ontario
  - Toronto Immune & Digestive Health Institute /ID# 274259, Toronto, Ontario
  - Diex Recherche Quebec Inc. /ID# 274268, Québec
- China (16):
  - The First Affiliated Hospital Of Anhui Medical University /ID# 274786, Hefei, Anhui
  - Chongqing General Hospital /ID# 274564, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital, Sun-Yat Sen University /ID# 274823, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 274843, Guangzhou, Guangdong
  - The Second Hospital Of Hebei Medical University /ID# 274822, Shijiazhuang, Hebei
  - The Second Affiliated Hospital Of Zhengzhou University /ID# 274569, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 274563, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 274616, Wuhan, Hubei
  - The Second Xiangya Hospital Of Central South University /ID# 274712, Changsha, Hunan
  - Nanjing Drum Tower Hospital /ID# 274710, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 274801, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 274784, Changchun, Jilin
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 275658, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University /ID# 275478, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 274849, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine /ID# 274689, Hangzhou, Zhejiang
- Croatia (5):
  - Klinicki Bolnicki Centar Zagreb /ID# 273316, Grad Zagreb, City of Zagreb
  - Poliklinika Solmed /ID# 273323, Zagreb, City of Zagreb
  - Poliklinika Borzan d.o.o. /ID# 273324, Osijek, County of Osijek-Baranja
  - Specialty Hospital Medico /ID# 273334, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 273327, Split, Split-Dalmatia County
- Czechia (2):
  - Hepato-Gastroenterologie HK /ID# 276654, Hradec Králové, Hradec Kralove
  - Nemocnice Ceske Budejovice /ID# 276530, České Budějovice
- Estonia (3):
  - Parnu Hospital /ID# 273584, Pärnu
  - East Tallinn Central Hospital /ID# 273723, Tallinn
  - West Tallinn Central Hospital /ID# 273722, Tallinn
- Finland (2):
  - Kuopion Yliopistollinen Sairaala /ID# 274856, Kuopio, Northern Savonia
  - Turku University Hospital /ID# 274312, Turku, Southwest Finland
- France (5):
  - Chu de Nice-Hopital Larchet Ii /Id# 278595, Nice, Alpes-Maritimes
  - CHU de Montpellier - Hopital Saint Eloi /ID# 278594, Montpellier, Herault
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 278633, Créteil, Paris
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 278587, St-Priest-en-Jarez, Pays de la Loire Region
  - Hopital Saint Antoine /ID# 278593, Paris
- Germany (20):
  - Universitaetsklinikum Freiburg /ID# 274763, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 273411, Ulm, Baden-Wurttemberg
  - Medizinisches Versorgungszentrum Dachau /ID# 273458, Dachau, Bavaria
  - Universitaetsklinikum Erlangen /ID# 273504, Erlangen, Bavaria
  - Markus Krankenhaus /ID# 273436, Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt /ID# 273462, Frankfurt am Main, Hesse
  - Universitaetsmedizin Essen /ID# 273505, Essen, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 273447, Minden, North Rhine-Westphalia
  - Magen-Darm-Zentrum-Remscheid /ID# 273435, Remscheid, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 273448, Dresden, Saxony
  - Eugastro /ID# 273573, Leipzig, Saxony
  - Studiengesellschaft BSF Unternehmergesellschaft /ID# 273457, Halle, Saxony-Anhalt
  - Praxisgemeinschaft Jerichow Schulze /ID# 273433, Jerichow, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel /ID# 273463, Kiel, Schleswig-Holstein
  - Praxis fuer Gastroenterologie /ID# 274546, Lübeck, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 274545, Berlin
  - Drk Kliniken Berlin - Köpenick /ID# 273514, Berlin
  - Krankenhaus Waldfriede /ID# 273708, Berlin
  - GSGH Gastroenterologische Studiengesellschaft Herne GbR /ID# 273459, Herne
  - Universitaetsklinikum Regensburg /ID# 273519, Regensburg
- Hungary (9):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 275083, Debrecen, Hajdú-Bihar
  - Clinfan /ID# 274904, Szekszárd, Tolna County
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 275077, Szombathely, Vas County
  - Obudai Egeszsegugyi Centrum /ID# 274919, Budapest
  - Eszak-Pesti Centrumkorhaz - Honvedkorhaz - Podmaniczky Utca /ID# 275722, Budapest
  - Semmelweis Egyetem /ID# 274872, Budapest
  - Semmelweis Egyetem /ID# 274883, Budapest
  - Pannónia Magánorvosi Centrum /ID# 275723, Budapest
  - Szegedi Tudomanyegyetem /ID# 275185, Szeged
- Ireland (6):
  - Portiuncula University Hospital /ID# 273782, Ballinasloe, Galway
  - Our Lady of Lourdes Hospital - Drogheda /ID# 273783, Drogheda, Louth
  - Midland Regional Hospital Mullingar /ID# 273784, Mullingar, Westmeath
  - St. Vincent's University Hospital /ID# 274617, Dublin
  - Beaumont Hospital /ID# 273787, Dublin
  - Connolly Hospital /ID# 274173, Dublin
- Israel (6):
  - Yitzhak Shamir Medical Center /ID# 275525, Ẕerifin, Central District
  - Assuta Ashdod Medical Center /ID# 274686, Ashdod, Southern District
  - Soroka Medical Center /ID# 273350, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 273348, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 273351, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus- Haifa /ID# 273347, Haifa
- Italy (10):
  - Azienda Ospedaliero Universitaria di Cagliari - P.O. Duilio Casula /ID# 274683, Monserrato, Cagliari
  - IRCCS Istituto Clinico Humanitas /ID# 274518, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 274516, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 274828, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 274685, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 274520, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 274517, Milan
  - Azienda Ospedale-Universita Padova /ID# 274519, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 274824, Palermo
  - Azienda Ospedaliero Universitaria Pisana /ID# 274829, Pisa
- Latvia (3):
  - Liepaja Regional Hospital /ID# 275164, Liepāja
  - Pauls Stradins Clinical University Hospital /ID# 273586, Riga
  - Digestive Diseases Center GASTRO /ID# 273589, Riga
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 273590, Kaunas
  - Panevezys Republican Hospital /ID# 273592, Panevezys
  - Vilnius University Hospital Santaros Klinikos /ID# 273591, Vilnius
  - Inlita - Lazdynai CTC /ID# 273725, Vilnius
- Netherlands (6):
  - Radboudumc /ID# 274797, Nijmegen, Gelderland
  - Elisabeth TweeSteden Ziekenhuis /ID# 274940, Tilburg, North Brabant
  - OLVG - Locatie Oost /ID# 274809, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC /ID# 274939, Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk /ID# 274936, Dordrecht, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis /ID# 274806, Rotterdam, South Holland
- Poland (10):
  - RIVERMED Sp. z o. o. /ID# 274420, Poznan, Greater Poland Voivodeship
  - Osrodek Badan Klinicznych Clinsante /ID# 274190, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - PROMED P. Lach, R. Glowacki S.j /ID# 274392, Krakow, Lesser Poland Voivodeship
  - EMC Instytut Medyczny S.A /ID# 275113, Wroclaw, Lower Silesian Voivodeship
  - Centrum Zdrowia Mdm /ID# 274192, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA /ID# 274538, Warsaw, Masovian Voivodeship
  - WSD MEDI Clinical Sp. z o.o. /ID# 274194, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Lukamed Sp. z o.o /ID# 274193, Chojnice, Pomeranian Voivodeship
  - Novamed Robert Koteras /ID# 274547, Bytom, Silesian Voivodeship
  - Twoja Przychodnia Szczecińskie Centrum Medyczne /ID# 274187, Szczecin, West Pomeranian Voivodeship
- Puerto Rico (3):
  - Isis Clinical Res. Ctr P.S.C. /ID# 274859, Guaynabo
  - CMRC Headlands LLC /ID# 274832, San Juan
  - Fdi Clinical Research /ID# 275337, San Juan
- Romania (5):
  - Memorial Healthcare International S.R.L. /Id# 276040, Bucharest, București
  - Spitalul Clinic Colentina /ID# 275892, Bucharest, București
  - Clinica Gastro Med SRL /ID# 275891, Cluj-Napoca, Cluj
  - OncoHelp Association /ID# 275889, Timișoara, Timiș County
  - Monza-Ares S.R.L. /Id# 276048, Bucharest
- Saudi Arabia (3):
  - King Saud University /ID# 274818, Riyadh, Riyadh Region
  - King Faisal Specialist Hospital and Research Center /ID# 274819, Riyadh, Riyadh Region
  - King Fahad Specialist Hospital /ID# 274820, Dammam
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 274740, Banská Bystrica, Banská Bystrica Region
  - ENDOMED s.r.o /ID# 274734, Košice
- Slovenia (2):
  - General Hospital Celje /ID# 275127, Celje
  - University Medical Centre Ljubljana /ID# 273636, Ljubljana
- South Korea (10):
  - Inje University Haeundae Paik Hospital /ID# 274435, Busan, Busan Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 274439, Daegu, Daegu Gwang Yeogsi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 274429, Daejeon, Daejeon Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 274441, Seongnam-si, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 274433, Suwon, Gyeonggido
  - Chosun University Hospital /ID# 276672, Gwangju, Jeonranamdo
  - Seoul National University Hospital /ID# 274438, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 274431, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital /ID# 274436, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 274440, Seoul, Seoul Teugbyeolsi
- Spain (12):
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 274266, Santiago de Compostela, A Coruna
  - Hospital General De Granollers /ID# 274384, Granollers, Barcelona
  - Sant Joan de Deu de Manresa /ID# 274288, Manresa, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrín /ID# 274277, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundación Alcorcón /ID# 274309, Alcorcón, Madrid
  - Hospital Universitario Puerta De Hierro /ID# 274271, Majadahonda, Madrid
  - Hospital de Cabueñes /ID# 274254, Gijón, Principality of Asturias
  - Hospital Universitario Virgen Macarena /ID# 274258, Seville, Sevilla
  - Hospital Clinic de Barcelona /ID# 274262, Barcelona
  - Complejo Hospitalario Universitario de Pontevedra /ID# 274269, Pontevedra
  - Consorci Hospital General Universitario de Valencia /ID# 274275, Valencia
  - Hospital Universitario Doctor Peset /ID# 274385, Valencia
- Sweden (5):
  - Danderyds Sjukhus - Danderyd /ID# 274401, Danderyd, Stockholm County
  - Karolinska University Hospital Solna /ID# 274379, Solna, Stockholm County
  - Alingsås Lasarett /ID# 274399, Alingsås, Västra Götaland County
  - Universitetssjukhuset Örebro /ID# 274386, Örebro, Örebro County
  - Linkoping University Hospital /ID# 274932, Linköping, Östergötland County
- Switzerland (3):
  - Luzern Kantonsspital /ID# 275415, Lucerne, Canton of Lucerne
  - Kantonsspital St.Gallen /ID# 273382, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Universitaetsspital Bern /ID# 273364, Bern
- Taiwan (5):
  - China Medical University Hospital /ID# 273641, Taichung
  - National Taiwan University Hospital /ID# 273632, Taipei
  - Mackay Memorial Hospital /ID# 273643, Taipei
  - Taipei Veterans General Hospital /ID# 274717, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 273640, Taoyuan
- United Arab Emirates (3):
  - Burjeel Medical City /ID# 274749, Abu Dhabi
  - Sheikh Shakhbout Medical City /ID# 274643, Abu Dhabi
  - Sheikh Khalifa Medical City /ID# 274777, Abu Dhabi
- United Kingdom (8):
  - Barts Health NHS Trust - The Royal London Hospital /ID# 274959, London, Greater London
  - King'S College Hospital /ID# 275223, London, Greater London
  - Velocity North London /ID# 275581, North Finchley, Greater London
  - Queen Elizabeth University Hospital - NHS Greater Glasgow and Clyde /ID# 274758, Glasgow, Lanarkshire
  - Fairfield General Hospital /ID# 274947, Manchester, Lancashire
  - The John Radcliffe Hospital /ID# 274757, Oxford, Oxfordshire
  - Queen Elizabeth Hospital Birmingham /ID# 275287, Birmingham
  - Stepping Hill Hospital-Stockport NHS foundation trust /ID# 275838, Stockport

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-540